CLINICAL TRIAL: NCT00366574
Title: Comparison of INTRALASE® to AMADEUS™ Microkeratome
Brief Title: Comparison of a Laser Keratome to a Mechanical Microkeratome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-05-003
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2005-03

CONDITIONS: Myopia; Astigmatism; Myopic Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

INTERVENTIONS:
Device: Amadeus Microkeratome
Device: IntraLase

SUMMARY:
The purpose of this study was to evaluate the performance of the INTRALASE®, a laser keratome which creates a corneal flap, and compare it to a mechanical microkeratome (Amadeus™). Our hypothesis is that there is no difference between the 2 devices.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for bilateral wavefront-guided LASIK
* Myopia up to -7.00 D
* Astigmatism of 0.00 to -1.50 D

Exclusion Criteria:

* History of ocular pathology
* Previous ocular surgery
* Very large pupils (greater than 8mm diameter, infrared measurement)
* Thin corneas (preoperatively calculated minimal residual bed < 250 um)
* Irregular astigmatism
* Asymmetric astigmatism
* Unstable refraction
* Any other criteria that precludes subject to undergo LASIK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-09; Study Completion 2005-02

PRIMARY OUTCOMES:
Visual acuity
Contrast sensitivity
Induction of high order aberration
Corneal sensation

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Medical University of South Carolina